CLINICAL TRIAL: NCT00224094
Title: A Comparison of Transdermal vs. Oral Estrogen Replacement Therapy on Androgen Levels and Thyroid Function in Naturally Menopausal Women
Brief Title: A Comparison of Patch vs. Pill Estrogen Therapy on Testosterone Levels and Thyroid Tests in Menopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ALO0102
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Menopause
Keywords: Menopause; Testosterone; Androgens; Sex Hormone Binding Globulin; Thyroid function; Cortisol
MeSH Terms: interventions — Estrogens, Conjugated (USP); Administration, Cutaneous

ARMS (2):
- Sequence A (Experimental): Oral ERT then transdermal ERT
  Interventions: Drug: Premarin® (oral) vs. Alora® (transdermal)
- Sequence B (Experimental): Transdermal ERT then oral ERT
  Interventions: Drug: Premarin® (oral) vs. Alora® (transdermal)

INTERVENTIONS:
Drug: Premarin® (oral) vs. Alora® (transdermal)

SUMMARY:
This study compares the effects of 12 weeks of treatment with transdermal versus oral estrogen therapy on testsoterone levels and thyroid tests in healthy, naturally menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Naturally menopausal women
* Aged 42-70 years
* Currently using combination estrogen-progestin replacement therapy

Exclusion Criteria:

* Women with contraindications to HRT use, including:Unexplained vaginal bleeding, liver disease, breast or endometrial cancer, venous thromboembolic events
* Thyroid disease
* Adrenal disease

Ages: 42 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2002-01; Primary Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Compare the effects of a 12-week course of oral CEE to a 12-week course of transdermal estradiol on free testosterone concentrations in menopausal women. | 12 weeks

SECONDARY OUTCOMES:
Compare the effects of oral versus transdermal ERT on thyroid binding globulin concentrations and tests of thyroid function. | 12 weeks
Compare the effects of oral versus transdermal ERT on cortisol binding globulin and total and free cortisol concentrations. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jan L Shifren, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States